CLINICAL TRIAL: NCT06843629
Title: Clinical Application of PET Imaging Targeting MSLN in Malignant Tumors
Status: Recruiting | Type: Observational
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Other Study IDs: Wuhan Union Hospital, China
Record Dates: First submitted 2024-12-20; First posted 2025-02-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2024-10

CONDITIONS: Ovarian Cancer; Lung Adenocarcinoma; Pancreatic Cancer
MeSH Terms: conditions — Ovarian Neoplasms; Adenocarcinoma of Lung; Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Specific positron imaging agents targeting MSLN — To perform integrated PET/MR or PET/CT visualization of patients with clinically suspected or confirmed pancreatic cancer, ovarian cancer, lung adenocarcinoma and other malignant tumors with high MSLN expression and healthy volunteers, using specific positron imaging agents targeting MSLN (taking [68Ga]Ga-NOTA-MSLN antibody fragment as an example), to achieve the following purposes: Patients with malignant tumors: for diagnosis and staging of diseases, comparing with the gold standard pathological diagnosis, evaluating diagnostic efficacy, clarifying the presence or absence of lesions, and determining the location and nature of lesions; comparing with [18F]FDG PET for accurate staging, evaluating the tumor load, and helping to determine the therapeutic plan. Healthy volunteers: Pharmacokinetic analysis will be performed to clarify the distribution and metabolism of the drug in the body and its safety.

SUMMARY:
The project aims to perform integrated PET/MR or PET/CT visualization of patients with clinically suspected or confirmed pancreatic cancer, ovarian cancer, lung adenocarcinoma and other malignant tumors with high MSLN expression and healthy volunteers, using targeted MSLN-specific imaging agents (taking [68Ga]Ga-NOTA-MSLN antibody fragment as an example), to achieve the following purposes: Patients with malignant tumors: for diagnosis and staging of diseases, comparing with the gold standard pathological diagnosis, evaluating diagnostic efficacy, clarifying the presence or absence of lesions, and determining the location and nature of lesions; comparing with [18F]FDG PET for accurate staging, evaluating the tumor load, and helping to determine the therapeutic plan. Healthy volunteers: Pharmacokinetic analysis will be performed to clarify the distribution and metabolism of the drug in the body and its safety.

DETAILED DESCRIPTION:
Malignant tumors are a major public health problem affecting global health. According to Globocan data, in 2020, there will be about 19.3 million new cases of malignant tumors and 9.9 million deaths worldwide. In China, there will be about 1.56 million new cases and 910,000 deaths, ranking first in the world. The global burden of disease is dominated by the burden of cancer, which will continue to increase globally for at least the next 20 years. However, in the early stages, most cancers are largely asymptomatic or have only a few nonspecific symptoms, including fever, nausea, vomiting, changes in stool characteristics, cough, etc., which are often overlooked, and therefore, exploring new strategies for the early and accurate diagnosis of malignant tumors has a crucial role to play in improving the prognosis of patients. Mesothelin (MSLN) is a glycosylphosphatidylinositol-anchored protein that is expressed at low levels in healthy mesothelial tissues (pleura, peritoneum, pericardium) but appears to be highly expressed in many cancer cells, especially in cancers characterized by invasiveness and poor prognosis, including pancreatic, ovarian, and lung adenocarcinomas. Preclinical studies have shown that MSLN expression has a positive role in malignant transformation and chemoresistance through the Wnt/NF-κB/ERK1/2/Akt signaling pathway. Abnormal expression of MSLN plays an important role in tumor cell growth, invasion and metastasis. Meanwhile, MSLN overexpression can activate the PI3K pathway and induce drug resistance in pancreatic cancer cells. In addition, MSLN has become a popular target for targeted antitumor therapy due to its high differential expression, including monoclonal antibodies, antibody drug combinations (ADCs), radioimmunotherapy (RIT), and CAR-T cellular immunotherapy for mesothelioma. Several antibody-drug conjugates (ADCs) against MSLN have been developed, such as LMB-100 (also known as RG7787) as an antibody-drug coupling targeting MSLN, which has been effective in terms of efficacy.Haas et al. utilized lentiviral transduction of chimeric antigen receptor (CAR)-modified autologous T-cells to target anti-MSLN in patients with malignant pleural mesothelioma, ovarian cancer and pancreatic cancer patients, and the results proved to be safe and feasible. Therefore, MSLN is an important target for precise diagnosis and treatment of malignant tumors.

Currently, high-quality, accurate imaging, multiphase computed tomography (CT) and magnetic resonance imaging (MRI) are widely used for detection, staging, and treatment planning. However, CT and MRI scans frequently detect lesions that cannot be further defined, and enhanced CT and enhanced MR also remain limited to morphological features of the tumor. This leads to uncertainty in the diagnosis or extent of disease. For example, overlapping imaging of adenocarcinoma of the pancreas and chronic pancreatitis has led to an indistinguishable misdiagnosis rate of up to 25%. Although endoscopic retrograde cholangiography and cholangiography may provide additional evidence of inflammatory etiology rather than malignancy, these methods are invasive, carry the risk of tumor dissemination along the needle tracks, and may also have a false-negative rate of up to 60%. FDG is a nonspecific tumor imaging agent. Because the energy metabolism of lymphocytes, monocytes, and other inflammatory cells during phagocytosis is also dominated by anaerobic glycolysis, proliferative lesions such as infections and granulomas, and nonmalignant lesions such as benign tumors, may also show high uptake of [18F]FDG. False-positive PET/CT cases are mainly inflammatory lesions of the pancreas (autoimmune pancreatitis, chronic pancreatitis), and granulomatous lesions (pancreatic tuberculosis). Compared with the conventional imaging agent [18F]FDG. 68Ga-labeled Fibroblast Activation Protein (FAP) inhibitors have higher uptake in tumor and lower uptake in other normal tissues, resulting in a higher Target-to-Background Ratio (TBR), which is conducive to improving their sensitivity in detecting tumor. However, 68Ga-FAPI-04 is not a tumor-specific imaging agent, and fibrosis caused by some other benign lesions may also lead to increased FAP expression. Xiaoli Lan, Kirienko M et al. showed that FAP is also expressed in pancreatic α-cells, which is another important factor limiting the use of 68Ga-FAPI-04 in the diagnosis of pancreatic cancer. With the growth of MSLN-targeted therapies in the field of oncology, the development of MSLN-targeted PET imaging strategies as companion diagnostics will hopefully optimize MSLN-targeted therapies. Lamberts LE et al. used 89Zr-MMOT0530A PET to visualize pancreatic and ovarian cancer lesions and antibody biodistribution, a technique that could potentially guide personalized antibody-based therapy. Linda N. Broer's study revealed the potential of 89Zr-MSLN PET to respond to MSLN expression and 227Th-MSLN tumor uptake and biodistribution, demonstrating the potential of 89Zr-MSLN PET as a tool for predicting 227Th-MSLN antitumor activity. Hou's study revealed that the 124I-anti-MSLN probe demonstrated a rapid metabolic rate and the ability to specifically identify MSLN-positive tumors in vivo.

To sum up, this project carries out integrated PET/MR or PET/CT visualization of patients with clinically suspected or diagnosed pancreatic cancer, ovarian cancer, lung adenocarcinoma and other malignant tumors with high expression of MSLN and healthy volunteers, using targeted MSLN-specific imaging agents ([68Ga]Ga-NOTA-MSLN antibody fragment for example), with a view to achieving the following purposes: (1) Patients with malignant tumors: for diagnosis and staging of diseases, comparing with the gold standard pathological diagnosis, assessing diagnostic efficacy, clarifying the presence or absence of lesions, and judging the location and nature of lesions; comparing with [18F]FDG PET for accurate staging, evaluating the tumor load, and helping to determine the treatment plan. (2) Healthy volunteers: Pharmacokinetic analysis will be performed to clarify the metabolic pattern and adverse reactions of the drug in the body.

ELIGIBILITY:
Inclusion Criteria:

* Each subject must meet all enrollment criteria to be eligible to participate in the study:

  1. The subject or his/her legal representative is able to sign and date the informed consent form;
  2. A commitment to comply with the research procedures and to cooperate in the implementation of the full research process;
  3. Adult patients or healthy volunteers (aged 18 or above) of either sex;
  4. Patients with clinically suspected or confirmed malignant tumors such as pancreatic cancer, ovarian cancer, or lung adenocarcinoma (supporting evidence includes serum-related tumor markers, imaging data such as ultrasound, CT, MRI, etc., and histological pathology examination, etc.) and in good general condition;
  5. Consistent with the results of specific laboratory tests;
  6. Females of childbearing potential who have been using contraception for at least one month prior to screening and who are committed to using contraception for the entire study period and until a specified time after the end of the study；
  7. Other set entry criteria.

Exclusion Criteria:

* All subjects who meet any of the exclusion criteria baseline will be excluded from the study:

  1. Those who are unable to complete a PET/MR or PET/CT examination (including inability to lie down, claustrophobia, radiophobia, etc.);
  2. Having other comorbidities;
  3. Patients with known hypersensitivity to MSLN antibody fragment developers or synthetic excipients; fasting blood glucose level greater than 11.0 mmol/L prior to 18F-FDG injection；
  4. Have a history of comorbid drug use;
  5. Patients considered by the investigator to have poor compliance;
  6. Patients during pregnancy or lactation;
  7. Persons with other factors that make participation in this test inappropriate.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with clinically suspected or confirmed malignant tumors such as pancreatic cancer, ovarian cancer, or lung adenocarcinoma (supporting evidence includes serum-related tumor markers, imaging data such as ultrasound, CT, MRI, etc., and histological pathology examination, etc.) who are in good general condition.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Visual and standardized uptake values assessment of lesions and biodistribution | 1 year
  At least two experienced nuclear medicine physicians will conduct a visual analysis using consensus reading. The standardized uptake value (SUV) of tumor and organs will be measured after a semiquantitative analysis is conducted for each case. The SUV ranges from 0 to infinity, and a higher score means a higher uptake of targeting MSLN nuclear probe by the tumor, which implies a greater threat of the tumor being malignant or higher stage.

SECONDARY OUTCOMES:
Radioactivity in the blood and urine samples | 1 year
  Blood samples were collected at 25 minutes, 55 minutes and 115 minutes after injection.
Pathological sections of tumour tissue | 1 year
  The excised tumour tissue was taken for immunohistochemistry to verify its MSLN expression

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoli Lan, PhD, Study Director — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Wuhan Union Hospital, China, Wuhan, Hubei, China